CLINICAL TRIAL: NCT03794349
Title: A Phase 2 Randomized Study of Irinotecan/Temozolomide/Dinutuximab With or Without Eflornithine (DFMO) in Children With Relapsed, Refractory or Progressive Neuroblastoma
Brief Title: Irinotecan Hydrochloride, Temozolomide, and Dinutuximab With or Without Eflornithine in Treating Patients With Relapsed or Refractory Neuroblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL1821; NCI-2018-03377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL1821 (Other: Children's Oncology Group); ANBL1821 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: High Risk Neuroblastoma; Recurrent Neuroblastoma; Refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Eflornithine; Irinotecan; sargramostim; Colony-Stimulating Factors; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (chemotherapy, dinutuximab, sargramostim) (Active Comparator): Patients receive temozolomide PO, via NG, or G tube on days 1-5, irinotecan hydrochloride IV over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC or IV over 2 hours on days 6-12 of a 21-day cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dinutuximab; Drug: Irinotecan Hydrochloride; Biological: Sargramostim; Drug: Temozolomide
- Regimen B (eflornithine, chemotherapy, dinutuximab) (Experimental): Patients receive eflornithine PO, via NG, or G tube on days -6 to 7 and days 15-21 of cycle 1 and days 1-7 and 15-21 of subsequent cycles, temozolomide PO, via NG, or G tube on days 1-5, irinotecan hydrochloride IV over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC or IV over 2 hours on days 6-12. Treatment duration is 28 days for cycle 1 and then every 21 days in subsequent cycles for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dinutuximab; Drug: Eflornithine Hydrochloride; Drug: Irinotecan Hydrochloride; Biological: Sargramostim; Drug: Temozolomide

INTERVENTIONS:
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Drug: Eflornithine Hydrochloride — Given PO or via NG or G tube
  Other Names: alpha-Difluoromethylornithine hydrochloride; Eflornithine.HCl; Iwilfin; MDL 71782; MDL-71782; MDL71782; Ornidyl; RMI 71782; RMI-71782; RMI71782; Vaniqa
  Arms: Regimen B (eflornithine, chemotherapy, dinutuximab)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Biological: Sargramostim — Given SC or IV
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Drug: Temozolomide — Given PO or via NG or G tube
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies how well irinotecan hydrochloride, temozolomide, and dinutuximab work with or without eflornithine in treating patients with neuroblastoma that has come back (relapsed) or that isn't responding to treatment (refractory). Drugs used in chemotherapy, such as irinotecan hydrochloride and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as dinutuximab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Eflornithine blocks the production of chemicals called polyamines that are important in the growth of cancer cells. Giving eflornithine with irinotecan hydrochloride, temozolomide, and dinutuximab, may work better in treating patients with relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether administration of eflornithine hydrochloride (eflornithine [DFMO]) in combination with dinutuximab, irinotecan hydrochloride (irinotecan) and temozolomide results in an improved response rate compared to dinutuximab, irinotecan and temozolomide in patients with relapsed or refractory neuroblastoma and therefore is a therapeutic regimen worthy of further testing in patients with newly-diagnosed high-risk neuroblastoma.

SECONDARY OBJECTIVES:

I. To compare progression-free survival and overall survival between patients receiving dinutuximab, irinotecan and temozolomide with and without the addition of DFMO.

II. To define the toxicity profile of DFMO administered with dinutuximab, irinotecan and temozolomide.

EXPLORATORY OBJECTIVES:

I. To characterize the immune and cytokine profiles of patients treated with DFMO/chemotherapy/dinutuximab combination and correlate with response to therapy.

II. To evaluate GD2 levels in tumor cells from patient bone marrow samples and correlate with response to therapy.

III. To explore whether the addition of DFMO to the dinutuximab and chemotherapy backbone affects pain as determined by patient report and opiate usage.

OUTLINE: Patients are randomized to 1 of 2 regimens.

REGIMEN A: Patients receive temozolomide orally (PO), via nasogastric (NG), or gastric (G) tube on days 1-5, irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim subcutaneously (SC) or IV over 2 hours on days 6-12 of a 21-day cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

REGIMEN B: Patients receive eflornithine PO, via NG, or G tube on days -6 to 7 and days 15-21 of cycle 1 and days 1-7 and 15-21 of subsequent cycles, temozolomide PO, via NG, or G tube on days 1-5, irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC or IV over 2 hours on days 6-12. Treatment lasts 28 days for cycle 1 and then every 21 days for subsequent cycles up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of neuroblastoma or ganglioneuroblastoma or demonstration of neuroblastoma cells in the bone marrow with elevated urinary catecholamines (i.e. > 2 x upper limit of normal [ULN]), at the time of initial diagnosis.
* For the purposes of this study, aggressive multidrug chemotherapy is defined as chemotherapy including 2 or more agents that must include an alkylating agent and a platinum-containing compound as intended to treat high-risk disease. The doses of chemotherapy must be comparable to those used in frontline high-risk neuroblastoma therapies (examples include A3973, ANBL0532, ANBL09P1, ANBL12P1, and ANBL1531). Patients must have ONE of the following:

  * First episode of recurrent high-risk disease following completion of aggressive multi-drug frontline high-risk therapy.
  * First episode of progressive high-risk disease during aggressive multi-drug frontline therapy.
  * Primary resistant/refractory disease (less than partial response by International Neuroblastoma Response Criteria [INRC]) detected at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocol (examples include A3973, ANBL0532, ANBL09P1, ANBL12P1, ANBL1531, etc.).
* Patients must have at least ONE of the following at the time of enrollment:

  * Measurable tumor on magnetic resonance imaging (MRI) or computed tomography (CT) scan. Measurable is defined as >= 10 mm in at least one dimension on spiral/helical CT that is metaiodobenzylguanidine (MIBG) avid or demonstrates increased fludeoxyglucose F-18 (FDG) uptake on positron emission tomography (PET) scan.
  * MIBG-avid lesion detected on MIBG scan with positive uptake at a minimum of one site. This site must represent disease recurrence after completion of therapy, progressive disease on therapy, or refractory disease during induction.
  * Patients with resistant/refractory soft tissue disease that is not MIBG avid or does not demonstrate increased FDG uptake on PET scan must undergo biopsy to document the presence of viable neuroblastoma. Biopsy is not required for patients who have a new site of soft tissue disease (radiographic evidence of disease progression) regardless of whether progression occurs while receiving therapy or after completion of therapy.
  * Patients with bone marrow disease only will be eligible if they have more than 5% disease involvement (documented neuroblastoma cells) in at least one sample from bilateral bone marrow biopsies.
  * Note: Patients with elevated catecholamines (i.e. > 2 x ULN) only are NOT eligible for this study.
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age.
* Primary refractory/resistant patients must have received at least 4 cycles of frontline high-risk chemotherapy. Frontline therapy may also have included surgery, chemotherapy, autologous stem cell transplantation (SCT) +/- MIBG, immunotherapy, radiotherapy, and retinoids but must NOT have received second line therapy for resistant/refractory, relapsed, or progressive disease. Patients who received intensified therapy for poor induction response or refractory disease (e.g. MIBG) will be considered to have received second line therapy and will not be eligible.
* At least 14 days must have elapsed since completion of myelosuppressive therapy.
* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent.
* Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1.
* No interim time prior to study entry is required following prior radiation therapy (RT) for non-target lesions. However, patients must not have received radiation for a minimum of 4 weeks prior to study entry at the site of any lesion that will be identified as a target lesion to measure tumor response. Lesions that have been previously radiated cannot be used as target lesions unless there is radiographic evidence of progression at the site following radiation or a biopsy done following radiation shows viable neuroblastoma. Palliative radiation while on study is not permitted.
* Patients are eligible >= 6 weeks after autologous stem cell transplants or stem cell infusions (including stem cell infusions given as supportive care following 131 I-MIBG therapy) as long as hematologic and other eligibility criteria have been met.
* Patients are eligible >= 6 weeks after therapeutic 131 I-MIBG provided that all other eligibility criteria are met.
* Subjects who have previously received anti-GD2 monoclonal antibodies with or without retinoids for biologic therapy are eligible unless they have had progressive disease while receiving prior anti-GD2 therapy or progressed/relapsed within 3 months of receiving anti-GD2 therapy. However, eligible patients may NOT have received anti-GD2 monoclonal antibodies in combination with chemotherapy.
* Subjects who have received autologous marrow infusions or autologous stem cell infusions that were purged using monoclonal antibody linked to beads are eligible.
* Subjects who have previously received DFMO are eligible for this study provided they have not had progressive disease while receiving DFMO or progressed/relapsed within 3 months of completing DFMO.
* Patients must not have received long-acting myeloid growth factors (e.g. pegfilgrastim) within 14 days of entry on this study. Seven days must have elapsed since administration of a short-acting myeloid growth factor.
* For patients with solid tumors (without marrow involvement) including status post SCT: peripheral absolute neutrophil count (ANC) >= 750/uL (within 7 days prior to enrollment).
* For patients with solid tumors (without marrow involvement) including status post SCT: platelet count >= 75,000/uL (transfusion independent) (within 7 days prior to enrollment).
* Patients known to have bone marrow involvement with neuroblastoma are eligible provided that minimum ANC and transfusion independent platelet count criteria are met (as above). However, these patients are not evaluable for hematological toxicity.
* Creatinine clearance or radioisotope GFR >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years (male 0.6 mg/dL, female 0.6 mg/dL)
  * 2 to < 6 years (male 0.8 mg/dL, female 0.8 mg/dL)
  * 6 to < 10 years (male 1 mg/dL, female 1 mg/dL)
  * 10 to < 13 years (male 1.2 mg/dL, female 1.2 mg/dL)
  * 13 to < 16 years (male 1.5 mg/dL, female 1.4 mg/dL)
  * >= 16 years (male 1.7 mg/dL, female 1.4 mg/dL) (within 7 days prior to enrollment).
* Total bilirubin =< 1.5 x ULN for age (within 7 days prior to enrollment).
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5.0 x ULN for age (=< 225 U/L). For the purpose of this study, the ULN for SGPT is 45 U/L (within 7 days prior to enrollment).
* Shortening fraction of >= 27% by echocardiography (ECHO) (within 7 days prior to enrollment).
* Ejection fraction of >= 50% by ECHO or gated radionuclide study (within 7 days prior to enrollment).
* No evidence of dyspnea at rest, no exercise intolerance, no chronic oxygen requirement, and room air pulse oximetry > 94% if there is a clinical indication for pulse oximetry. Normal pulmonary function tests in patients who are capable of cooperating with testing (including diffusion capacity of the lung for carbon monoxide [DLCO)] are required if there is a clinical indication for determination. For patients who do not have respiratory symptoms, full pulmonary function tests (PFTs) are NOT required.
* Patients with a history of central nervous system (CNS) disease must have no clinical or radiological evidence of active CNS disease at the time of study enrollment.
* Patients with seizure disorders may be enrolled if seizures are well controlled on anti-convulsants.
* CNS toxicity =< grade 2.

Exclusion Criteria:

* Men and women of childbearing potential and their partners must agree to use adequate contraception while enrolled on this study. Based on the established teratogenic potential of alkylating agents, pregnant women will be excluded from this study. Because of potential risks to breastfed infants due to drug metabolites that could be excreted in breast milk, female patients who are lactating must agree to stop breastfeeding or will otherwise be excluded from this study. Females of childbearing potential must have a negative pregnancy test to be eligible for this study.
* Patients with only elevated catecholamines (i.e. > 2 x ULN) are NOT eligible for this study.
* Patients must have been off pharmacologic doses of systemic steroids for at least 7 days prior to enrollment. Patients who require or are likely to require pharmacologic doses of systemic corticosteroids while receiving treatment on this study are ineligible. The only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product administration in order to avoid allergic transfusion reactions. The use of conventional doses of inhaled steroids for the treatment of asthma is permitted, as is the use of physiologic doses of steroids for patients with known adrenal insufficiency.

Patients on any other immunosuppressive medications (e.g. cyclosporine, tacrolimus) are not eligible.

* Patients must not have received prior treatment with irinotecan and temozolomide.
* Patients must not have received enzyme-inducing anticonvulsants including phenytoin, phenobarbital, or carbamazepine for at least 7 days prior to study enrollment. Patients receiving non-enzyme inducing anticonvulsants such as gabapentin, valproic acid, or levetiracetam will be eligible.
* Patients who have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment are not eligible.
* Patients must not have been diagnosed with myelodysplastic syndrome or with any malignancy other than neuroblastoma.
* Patients with symptoms of congestive heart failure are not eligible.
* Patients must not have >= grade 2 diarrhea.
* Patients who are unable to tolerate oral/nasogastric/gastrostomy medications will not be eligible for this trial. Additionally, patients with significant malabsorption will not be eligible for this trial.
* Patients must not have uncontrolled infection.
* Patients with a history of grade 4 allergic reactions to anti-GD2 antibodies or reactions that required permanent discontinuation of the anti-GD2 therapy are not eligible.
* Patients with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of study agents or to significantly increase the severity of the toxicities experienced from study treatment are not eligible.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-04-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Macy, Principal Investigator — Children's Oncology Group
Locations (145):
- United States (124):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (11):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

REFERENCES:
- [Derived] Hogarty MD, Ziegler DS, Franson A, Chi YY, Tsao-Wei D, Liu K, Vemu R, Gerner EW, Bruckheimer E, Shamirian A, Hasenauer B, Balis FM, Groshen S, Norris MD, Haber M, Park JR, Matthay KK, Marachelian A. Phase 1 study of high-dose DFMO, celecoxib, cyclophosphamide and topotecan for patients with relapsed neuroblastoma: a New Approaches to Neuroblastoma Therapy trial. Br J Cancer. 2024 Mar;130(5):788-797. doi: 10.1038/s41416-023-02525-2. Epub 2024 Jan 10. PMID 38200233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with high-risk neuroblastoma in first relapse, primary refractory, or primary progressive disease enrolled between 7/8/2019 and 9/30/2024 across all COG institutions.
Period: Overall Study
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
Started | 46 | 48
Completed | 13 | 16
Not Completed | 33 | 32
Not completed — Adverse Event | 2 | 3
Not completed — Death | 0 | 2
Not completed — Physician Decision | 10 | 8
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Ineligible | 2 | 1
Not completed — Refusal | 2 | 3
Not completed — Progressive Disease | 7 | 10
Not completed — Stable Disease after 6 Cycles | 4 | 1
Not completed — Did not meet criteria to start next treatment cycle within 21 days after planned start of next cycle | 4 | 1
Not completed — Repeat eligibility studies before start of protocol therapy outside required eligibility parameters | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab) | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43 | 48 | 91
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 5.36 [1.08 to 21.22] | 6.14 [2.03 to 16.04] | 5.72 [1.08 to 21.22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 26 | 23 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 33 | 31 | 64
  Unknown or Not Reported | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 23 | 25 | 48
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79
  Canada | 1 | 3 | 4
  Australia | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Responders are defined as patients who achieve a >= minor response (MR) per the International Neuroblastoma Response Criteria (INRC) as their best overall response by the end of 6 cycles. The response rate to treatment will be calculated among all eligible patients, including placement of a 95% confidence interval on the response rate.
Time Frame: After every 2 cycles, for a maximum of 6 cycles of treatment (each cycle is 21 days)
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
Number analyzed (Participants) | 44 | 47
percentage of patients | 63.6 [48.9 to 76.2] | 57.4 [43.3 to 70.5]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Kaplan-Meier method will be used to estimate progression-free survival (PFS). PFS time will be calculated from the time of randomization to the occurrence of relapse, progressive disease, or death. Patients without a PFS event will be censored at the time of last follow-up. 1-Year PFS is provided.
Time Frame: Up to 1 year
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
Number analyzed (Participants) | 44 | 47
percentage of patients | 66.9 [52.1 to 81.7] | 56.0 [41.4 to 70.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier method will be used to estimate overall survival (OS). OS time will be calculated from the time of randomization to the occurrence of death. Patients still alive will be censored at the time of last follow-up.1-Year OS is provided.
Time Frame: Up to 1 year
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
Number analyzed (Participants) | 44 | 47
percentage of patients | 88.2 [78.0 to 98.4] | 82.0 [70.6 to 93.4]

4. Secondary Outcome: Incidence of Adverse Events >= Grade 3 (Regimen B)
Description: The percentage of patients on Regimen B with at least one Grade 3 or higher toxicity will be calculated, assessed with Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 5 years
Population: All eligible patients
Measure: Number; unit: percentage of patients
Arm/Group | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
Number analyzed (Participants) | 47
percentage of patients | 93.6

5. Other Pre Specified Outcome: Immune and Cytokine Profiles
Description: Will be assessed by exploring the relationship between response (responder versus [vs.] non-responder) after 6 cycles on Regimen B with serum cytokine levels (IL1, IL6, tumor necrosis factor [TNF]-alpha, IFN-gamma, etc.), tumor resident immune cells (natural killer [NK] cells, tumor-associated macrophages [TAMS], tumor infiltrating lymphocyte [TILS]), and critical immune cell suppressing proteins (B7H3, PDL-1) using Fisher's exact test for categorical and Wilcoxon rank-sum test for continuous factors.
Time Frame: Up to 6 cycles
Reporting Status: Not Posted

6. Other Pre Specified Outcome: GD2 Levels in Tumor Cells From Bone Marrow Samples
Description: Will be correlated with response (responder vs. non-responder) after 6 cycles using Fisher's exact test for categorical and the Wilcoxon rank-sum test for continuous factors.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Patient Reported Pain and Opiate Usage
Description: The occurrence of pain on each regimen as reported by patient report and opiate use will be descriptively summarized. Descriptive and summary statistics will be used to describe the scores from the Faces Pain Scale-Revised during the dinutuximab infusion and on day 1 with irinotecan and temozolomide alone for each arm separately. Confidence intervals will be constructed for the mean and frequency estimates. The day 1 patient reported outcome data are expected to be similar between the 2 regimens, while differences during or after completion of treatment may be observed.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years after enrollment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab)
All-Cause Mortality (participants affected / at risk) | 13/44 | 19/47
Serious Adverse Events (participants affected / at risk) | 3/44 | 20/47
Other Adverse Events (participants affected / at risk) | 34/44 | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) (N=44) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab) (N=47)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 5
Disease progression (General disorders) | 0 | 1
Fever (General disorders) | 0 | 7
Malaise (General disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 6
Upper respiratory infection (Infections and infestations) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2
Urine output decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (Chemotherapy, Dinutuximab, Sargramostim) (N=44) | Regimen B (Eflornithine, Chemotherapy, Dinutuximab) (N=47)
Anemia (Blood and lymphatic system disorders) | 12 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 5
Optic nerve disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 5
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 3 | 5
Fever (General disorders) | 9 | 7
Flu like symptoms (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 14 | 6
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 2
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 4
Lung infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viremia (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 5
Blood bilirubin increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 18 | 19
Lymphocyte count increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 19 | 21
Platelet count decreased (Investigations) | 6 | 8
Urine output decreased (Investigations) | 1 | 1
Weight gain (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 17 | 13
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 9
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Irritability (Psychiatric disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 5 | 7
Hypotension (Vascular disorders) | 3 | 0
Lymphedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03794349/Prot_SAP_000.pdf